CLINICAL TRIAL: NCT02867202
Title: A Randomized Clinical Trial to Assess the Efficacy of Intrauterine Balloon Compared to Intrauterine Contraceptive Device Plus Foley Catheter in the Therapy for Uterine Adhesion After Hysteroscopic Adhesiolysis
Brief Title: Adjuvant Therapy for Intrauterine Adhesions Between Two Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Feng Lin, attending doctor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wenzhou MC
Record Dates: First submitted 2016-04-11; First posted 2016-08-15 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Asherman Syndrome
Keywords: intrauterine balloon; Intrauterine Device Plus Foley Balloon Catheter; Asherman Syndrome
MeSH Terms: conditions — Gynatresia | interventions — Intrauterine Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrauterine balloon (Experimental): The heart-shaped intrauterine balloon is designed to fit into the cavity of the uterus,and removed on the 7th day after surgery. And hysteroscopy was taken out again after two or three months to re-evaluate the uterine adhesions.
  Interventions: Device: Intrauterine balloon
- intrauterine device Plus Foley Catheter (Experimental): Intrauterine Contraceptive Device Plus Foley Catheter are inserted into the uterine after hysteroscopic adhesiolysis. Foley Catheter is removed after three days while intrauterine device is removed at the second hysteroscopy. Uterine adhesions are judged again at the second hysteroscopy.
  Interventions: Device: Intrauterine Contraceptive Device Plus Foley Catheter

INTERVENTIONS:
Device: Intrauterine balloon — After the completion of hysteroscopic adhesiolysis, intrauterine balloon was inserted and inflated with 3-5 mL normal saline which was removed after 1 week.
  Other Names: Cook balloon
  Arms: Intrauterine balloon
Device: Intrauterine Contraceptive Device Plus Foley Catheter — After the completion of hysteroscopic adhesiolysis, Intrauterine Contraceptive Device Plus Foley Catheter were inserted into the uterine cavity. Foley Catheter was removed after three days and Intrauterine Device was removed at the second time of hysteroscopy.
  Other Names: Intrauterine Device Plus Foley Catheter
  Arms: intrauterine device Plus Foley Catheter

SUMMARY:
This study was taken out to compare two mechanical devices (intrauterine balloon and Intrauterine Contraceptive Device Plus Foley Catheter) in the therapy for intrauterine adhesions after hysteroscopic adhesiolysis. Participates were assigned into two groups by randomly.

DETAILED DESCRIPTION:
Intrauterine balloon and Intrauterine Contraceptive Device Plus Foley Catheter are both effective in the therapy for intrauterine adhesion.

The Intrauterine Contraceptive Device Plus Foley Catheter are usually inserted into the uterine after hysteroscopic adhesiolysis. Foley Catheter is removed after three days while intrauterine device is removed two or three month later.

The heart-shaped intrauterine balloon is designed to fit into the cavity of the uterus, and usually removed on the 7th day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe intrauterine adhesion (AFS score ≥5）
* Agreement to have a second-look hysteroscopy
* no previous history of hysteroscopic adhesiolysis

Exclusion Criteria:

* Minimal adhesion (AFS score<5)
* Previous hysteroscopic adhesiolysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, MD, Principal Investigator — The 1st Affiliated Hospital of Wenzhou Medical University
Locations (1):
- the 1st Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin XN, Zhou F, Wei ML, Yang Y, Li Y, Li TC, Zhang SY. Randomized, controlled trial comparing the efficacy of intrauterine balloon and intrauterine contraceptive device in the prevention of adhesion reformation after hysteroscopic adhesiolysis. Fertil Steril. 2015 Jul;104(1):235-40. doi: 10.1016/j.fertnstert.2015.04.008. Epub 2015 Apr 30. PMID 25936237
- [Background] Johary J, Xue M, Zhu X, Xu D, Velu PP. Efficacy of estrogen therapy in patients with intrauterine adhesions: systematic review. J Minim Invasive Gynecol. 2014 Jan-Feb;21(1):44-54. doi: 10.1016/j.jmig.2013.07.018. Epub 2013 Aug 9. PMID 23933351
- [Background] Lin X, Wei M, Li TC, Huang Q, Huang D, Zhou F, Zhang S. A comparison of intrauterine balloon, intrauterine contraceptive device and hyaluronic acid gel in the prevention of adhesion reformation following hysteroscopic surgery for Asherman syndrome: a cohort study. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):512-6. doi: 10.1016/j.ejogrb.2013.07.018. Epub 2013 Aug 7. PMID 23932377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients were recruited from 1st affiliated hospital of Wenzhou Medical University.
  Inclusion criteria were as follows:1) women aged 18 to 45 years. 2) agreed to have second-look hysteroscopy. 3) moderate to severe intrauterine adhesion (AFS score ≥5)
Pre-assignment Details: 1. not meeting inclusion criteria
  2. declined to participate
Groups:
- Intrauterine Balloon: After the completion of hysteroscopic adhesiolysis, intrauterine balloon was inserted and inflated with 3-5 mL normal saline which was removed after 1 week. And hysteroscopy was taken out again after two or three menstrual cycles to evaluate the uterine adhesions.
- Intrauterine Contraceptive Device Plus Foley Catheter: Intrauterine Contraceptive Device Plus Foley Catheter are inserted into the uterine after a hysteroscopic adhesiolysis. Foley Catheter is removed after three days while IUD removed at the second hysteroscopy. Uterine adhesions were judged again at the second hysteroscopy.
Period: Overall Study
Arm/Group | Intrauterine Balloon | Intrauterine Contraceptive Device Plus Foley Catheter
Started | 83 | 88
Completed | 62 | 56
Not Completed | 21 | 32

BASELINE CHARACTERISTICS:
Groups:
- Intrauterine Balloon: After the completion of hysteroscopic adhesiolysis, intrauterine balloon was inserted and inflated with 3-5 mL normal saline which was removed after 1 week.And hysteroscopy was taken out again after two menstrual cycles to evaluate the uterine adhesions.
- IUD Plus Foley Catheter: Intrauterine Contraceptive Device Plus Foley Catheter are inserted into the uterine after a hysteroscopic adhesiolysis. Foley Catheter is removed after three days while IUD removed at the second hysteroscopy. Uterine adhesions were judged again at the second hysteroscopy.
- Total: Total of all reporting groups
Arm/Group | Intrauterine Balloon | IUD Plus Foley Catheter | Total
Number analyzed (Participants) | 62 | 56 | 118
Age, Continuous [Mean (Standard Deviation); unit: year] | 31.69 (5.268) | 32.63 (6.125) | 32.14 (5.685)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 56 | 118
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 56 | 118
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 62 | 56 | 118
Parity [Mean (Standard Deviation); unit: Births] | 0.484 (0.565) | 0.554 (0.536) | 0.517 (0.551)

OUTCOME MEASURES:

1. Primary Outcome: the AFS Score at Second-look Hysteroscopy
Description: The AFS score is based on the American Fertility Society (AFS) Classification of Intra-uterine adhesions( 1988 version)The total range of AFS score is from 0 to 12, and the higher the score is, the worse the outcome is.
Time Frame: 2 or 3 months after the surgery
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Intrauterine Balloon: The heart-shaped intrauterine balloon is designed to fit into the cavity of the uterus,and removed on the 7th day after surgery. And hysteroscopy was taken out again after two menstrual cycles to evaluate the uterine adhesions.
  Intrauterine balloon: After the completion of hysteroscopic adhesiolysis, intrauterine balloon was inserted and inflated with 3-5 mL normal saline which was removed after 1 week.
- Intrauterine Device Plus Foley Catheter: Intrauterine Contraceptive Device Plus Foley Catheter are inserted into the uterine after a hysteroscopic adhesiolysis. Foley Catheter is removed after three days while Intrauterine Device is removed at the second hysteroscopy. Uterine adhesions are judged again at the second hysteroscopy.
  Intrauterine Contraceptive Device Plus Foley Catheter: After the completion of hysteroscopic adhesiolysis, Intrauterine Contraceptive Device Plus Foley Catheter were inserted into the uterine cavity. Foley Catheter was removed after three days and Intrauterine Device was removed at the second time of hysteroscopy.
Arm/Group | Intrauterine Balloon | Intrauterine Device Plus Foley Catheter
Number analyzed (Participants) | 62 | 56
Units on a scale | 6.5 [1 to 10] | 8 [3 to 12]
Statistical Analysis 1: Comparison: Intrauterine Balloon vs Intrauterine Device Plus Foley Catheter; Data analysis was performed with SPSS version 22.0, using two-sided test, and a p value < 0.05 was considered statistically significant; Test type: Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months to 1 year
Description: Among 171 participants who were initially recruited, 18 were excluded from analysis; 8 patients declined to participate and 10 patients did not meet the inclusion criteria. 30 participants subsequently refused to undergo the second-look hysteroscopy, and 5 subjects were also excluded for protocol violation. 17 women in the study reported side effects. 15 subjects suffered from moderate to severe postoperative pain; 12in the COOK balloon stent group and 3 in the IUD plus Foley catheter group.
Arm/Group | Intrauterine Balloon | IUD Plus Foley Catheter
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/88
Other Adverse Events (participants affected / at risk) | 21/83 | 32/88
OTHER ADVERSE EVENTS (reported when occurring in more than 2.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrauterine Balloon (N=83) | IUD Plus Foley Catheter (N=88)
suffered from moderate to severe postoperative pain (Injury, poisoning and procedural complications) | 12 (12) | 3 (3)
refuse to have second-look hysteroscopy (Investigations) | 9 (9) | 21 (21) — excluded
Protocol violation (Investigations) | 3 (3) | 2 (2) — excluded
Declined to participate (Investigations) | 4 (4) | 4 (4) — excluded
Not meeting inclusion criteria (Investigations) | 5 (5) | 5 (5) — excluded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02867202/SAP_000.pdf
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02867202/Prot_001.pdf